CLINICAL TRIAL: NCT05757687
Title: Evaluation of the Safety, Tolerability and Efficacy the Omega System for the Treatment of Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia
Brief Title: Evaluation of the Safety, Tolerability, and Efficacy of the Omega System for the Treatment of LUTS Due to BPH
Acronym: Omega
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ProArc Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA-CP-22
Record Dates: First submitted 2023-02-15; First posted 2023-03-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-05

CONDITIONS: Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Omega procedure (Experimental)
  Interventions: Device: Omega device

INTERVENTIONS:
Device: Omega device — The ProArc Medical Omega system is a prostatic reshaping device. The Omega System is comprised of two main components: Omega Delivery Device and Omega Implant.
  The delivery system uses a diathermy electrode to perform a circular and superficial incision through the urethral wall into the prostate tissue, into which the arc-shaped permanent implant is placed. The implant is made up of commonly used surgical implantable nitinol material, coated with Parylene coating. The implant expands the obstructed area, reducing the fluid obstruction through the prostatic urethra.

SUMMARY:
This is a prospective, two-stage, multi-center, pilot clinical study to evaluate the safety/tolerability/efficacy of the Omega System device. The Omega arc-shaped implant is inserted by the Omega delivery system into the prostate tissue of subjects to relieve lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH). The study will first evaluate the Omega system on patients undergoing prostatectomy, which is not indicated for the device.

ELIGIBILITY:
Stage 1

Inclusion Criteria:

1. Male ≥50 years of age and ≤ 80 years old.
2. Will undergo planned prostatectomy.
3. Participant understands and is willing to the informed consent form.
4. Prostate Volume between 30cc and 80cc.
5. Prostate length ≥ 3cm

Exclusion Criteria:

1. Unable to comply with the clinical protocol.
2. Vulnerable population such as inmates or developmentally delayed individuals.
3. Any medical condition or treatment, which in the opinion of the investigator may interfere with the procedure, such as:

   * Patient with coagulopathy due to medications or congenital condition - inability to stop taking anticoagulants and/or antiplatelets for at least 3 days prior to the procedure or coumadin for at least 5 days prior to the procedure (low dose aspirin therapy is not prohibited).
   * Use of alpha-blockers within 2 weeks of pre-treatment (baseline) evaluation.
   * Use of 5-α-reductase inhibitors within 6 months of pre-treatment (baseline) evaluation.
4. American Society of Anesthesiologists score (ASA) > 3.
5. Previous prostate surgery such as: TURP, stent implantations, laser prostatectomy, hyperthermia or another invasive treatment to the prostate.
6. Presence of an artificial urinary sphincter or stent(s) in the urethra or prostate.
7. Other urethral conditions that may prevent insertion of Delivery Device into prostatic urethra.
8. Previous rectal surgery, other than hemorrhoidectomy
9. Current gross hematuria.
10. Known allergy to nickel or titanium or stainless steel.

Stage 2

Inclusion Criteria:

1. Male ≥50 years old.
2. Suspected symptomatic benign prostatic hyperplasia (BPH).
3. International Prostate Symptom Score (IPSS) >13.
4. Peak flow rate ≤ 12 ml/sec (with voided volume ≥ 125ml).
5. Participant understands and is willing to the informed consent form.
6. Prostate Volume between 30cc and 80cc.
7. Prostate length ≥ 3cm and ≤ 5cm

Exclusion Criteria:

1. Diagnosed or suspected prostate cancer. If suspected, prostate cancer must be ruled out.
2. Concomitant participation in another interventional study.
3. Unable to comply with the clinical protocol including all the follow-up requirements.
4. Vulnerable population such as inmates or developmentally delayed individuals.
5. Significant comorbidities which would affect study participation.
6. Any medical condition or treatment, which in the opinion of the investigator may interfere with the procedure ,such as:

   * Use of concomitant medications (e.g., anticholinergics, antispasmodics, or antidepressants) affecting bladder function.
   * Patient with coagulopathy due to medications or congenital condition - inability to stop taking anticoagulants and/or antiplatelets for at least 3 days prior to the procedure or coumadin for at least 5 days prior to the procedure; low dose aspirin therapy not prohibited.
   * Alpha-blockers within 2 weeks of pre-treatment (baseline) evaluation.
   * Taking 5-alpha reductase inhibitors (5-ARI) within 6 months (3 months for type II 5-ARI) of pre-treatment (baseline) evaluation unless evidence of same drug dose for at least 6 months with a stable voiding pattern (the drug dose should not be altered or discontinued throughout the study).
   * Patient is taking steroids. [Note: Patients approved for the trial who are using the above medications will continue using them after the trial, except for Alpha blockers.]
7. Previous prostate surgery such as: TURP, stent implantations, laser prostatectomy, hyperthermia or another invasive treatment to the prostate.
8. Compromised renal function due to obstructive uropathy.
9. Active Urinary Tract Infection (UTI).
10. Obstructive or protruding median lobe.
11. American Society of Anesthesiologists score (ASA) > 3.
12. Known neurogenic bladder or neurological disorders that might affect bladder or function.
13. Recent myocardial infarction (less than three months).
14. Concomitant bladder stones.
15. Current gross hematuria.
16. Active or history of epididymitis within the past 3 months.
17. Presence of an artificial urinary sphincter or stent(s) in the urethra or prostate.
18. Confirmed or suspected malignancy of bladder.
19. History or presence of strictures in the anterior urethra or bladder neck contracture or detrusor muscle spasms.
20. Other urethral conditions that may prevent insertion of Delivery Device into prostatic urethra.
21. Bacterial prostatitis within the last 12 months.
22. Previous rectal surgery, other than hemorrhoidectomy.
23. Current uncontrolled diabetes (i.e., hemoglobin A1c ≥ 9%).
24. Known allergy to nickel or titanium or stainless steel.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2026-01-03 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary Safety (Stage 1 and Stage 2) - Incidence and severity of procedural and device related adverse events. | 12 Months
  Incidence and severity of procedural and device related adverse events.
Primary Safety (Stage 2) - Incidence of post-operative catheterization after 7 days, up to 14 days. | 2 weeks
  Incidence of post-operative catheterization after 7 days, up to 14 days.
Efficacy (Stage 2) - Change in urinary related symptom | 3 Months
  Improvement in urinary related symptoms as evidenced by at least 30% decrease in International Prostate Symptom Score (A score of 0-7 indicates mild symptoms, 8-19 indicates moderate symptoms and 20-35 indicates severe symptoms)

SECONDARY OUTCOMES:
Functionality (Stage 1) - Location and orientation of Omega implant in the prostate before prostatectomy is as planned: Yes/No | Procedure day
  Evaluating whether the outcome of the Omega implant's location and orientation turned out as the surgeon planned prior to the Omega procedure.
Functionality (Stage 1) - Location and depth Omega incision in the excised prostate is as planned: Yes/No. | Procedure day
  Evaluating whether the Omega incision location and depth outcome turned out as the surgeon planned prior to the Omega procedure.
Usability (Stage 1 and Stage 2) - Evaluate the usability of the device and entire process | Procedure day
  Evaluate the usability of the device and the entire process using the usability questionnaire (The highest score of 60 indicates that the device is extremely user-friendly, while the lowest score of 12 indicates that the device is very difficult to use)
Efficacy (Stage 2) - Improvement in urinary related symptoms | 1 Months, 6 Months and 12 months
  Evaluate the improvement in urinary-related symptoms as evidenced by a decrease of at least 30% in the IPSS score. (A score of 0-7 indicates mild symptoms, 8-19 indicates moderate symptoms and 20-35 indicates severe symptoms)
Efficacy (Stage 2) - Improvement of peak urinary flow rate as evidenced by an increase of at least 25% in uroflowmetry Qmax | 1 Months, 3 Months, 6 Months and 12 months
Exploratory - Change in PSA compared to baseline | 1 Months, 6 Months and 12 Months
Exploratory - Change in sexual function assessments from screening to 3, 6 and 12 months using the International Index of Erectile Function (IIEF) and Male Sexual Health Questionnaire for Ejaculatory Function (MSHQ-EjD). | 3 Months, 6 Months and 12 months
  The IIEF-15 score ranges from 6 to 75 and is used to classify erectile dysfunction (ED).
  An MSHQ-EjD score of 20 indicates the absence of ejaculatory dysfunction, while a score of 0 indicates a high level of ejaculatory dysfunction.
Exploratory - Change in VAS pain score | Procedure day, 1-2 weeks and 1 month
  A VAS pain score of (0-1 mm) indicates no pain,(2-4 mm) - mild pain, (4-7 mm) - moderate pain, and (7-10 mm) - severe pain.
Exploratory - Change in post-void residual (PVR) test | 1 Months, 3 Months, 6 Months and 12 months
Exploratory - Incidence of inflammation, assessed by cystoscope | 6 months
Exploratory - Omega coverage assessed by cystoscope | 6 months
Exploratory - Change in the BPHII score from Baseline | 1 Months, 3 Months, 6 Months and 12 months
Incidence of repeat invasive treatment for Lower Urinary Tract Symptoms (LUTS) or increase in dosage or initiation of new medication to treat symptoms of BPH | 12 months
Incidence of Device removal | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank Mastandrea, Dr, Study Director — Board Member and Medical Director
Locations (5):
- Georgia (5):
  - N(N)LE New Vision University Hospital, Tbilisi
  - Israeli-Georgian Medical Research Clinic Healthycore, Tbilisi
  - JSC L.Managadze National Center of Urology, Tbilisi
  - Tbilisi Heart Center, Tbilisi
  - Todua Clinic, Tbilisi

IPD SHARING:
Plan to Share IPD: No